CLINICAL TRIAL: NCT01057758
Title: Effect of the Association of a Statin to Antibiotics on the Prognosis of Patients Presenting With a Suspicion of Ventilator-associated Pneumonia
Brief Title: STATIN-VAP STATIN-VAP - STATINs and Ventilator-Associated Pneumonia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: stopped for futility
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-002019-42; 2008 13 (Other: 2008 13)
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-04

CONDITIONS: Pneumonia
Keywords: Suspicion of ventilator-associated pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PLACEBO (Placebo Comparator): Half of the patients will be randomized to the placebo
  Interventions: Drug: PLACEBO
- Simvastatin (Active Comparator): Half of the subjects will receive the active drug, Simvastatin.
  Interventions: Drug: SIMVASTATIN

INTERVENTIONS:
Drug: SIMVASTATIN — Patients will receive 60 mg of study drug daily by mouth or feeding tube for 28 days or until discharged from the study ICU.
  Arms: Simvastatin
Drug: PLACEBO — Patients will receive one placebo by mouth or feeding tube daily for 28 days or until discharged form study ICU
  Arms: PLACEBO

SUMMARY:
The objective is to assess the efficacy and safety of oral simvastatin in patients with a suspicion of ventilator-associated pneumonia (VAP). The hypothesis of this study is that simvastatin therapy will improve mortality in patients a suspicion of VAP.

DETAILED DESCRIPTION:
When a patient will present a suspicion of VAP (Clinical Pulmonary Infection Score modified ≥ 5), Simvastatin or placebo will be administered with antibiotics. Quantitative cultures will be performed for microbiological confirmation of VAP. Simvastatin or placebo will be administered through an enteral feeding tube or administered orally when patients are able to safely take oral medications. The type and placement of the enteral feeding tube (nasogastric, nasoenteric, PEG, orogastric, oroenteric, etc.) and the ability to safely take oral medications will be determined by the patient's primary team. Study drug will be blinded with an identical appearing placebo.

Sequential Organ Failure Assessment score (SOFA), and various blood factors will be measured during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Duration of mechanical ventilation > 48 h
* First episode of suspicion of VAP with a Clinical Pulmonary Infection Score modified ≥ 5
* BAL, plugged telescopic catheter and/or tracheal aspirates quantitative cultures performed prior administration of antibiotics
* Informed consent

Exclusion Criteria:

* Statin treatment received under mechanical ventilation
* Age less than 18 years
* Pregnancy
* Unable to receive or unlikely to absorb enteral study drug
* Patient, surrogate, or physician not committed to full support ).
* Moribund patient with a SAPS II score > 75
* Simvastatin specific exclusions Allergy or intolerance to statins Physician insistence for the use or avoidance of statins during the current hospitalization CK , ALT or AST > 5 times the upper limit of normal Receiving cyclosporine, gemfibrozil, lopinavir, ritonavir itraconazole, kétoconazole, érythromycine, clarithromycine, télithromycine, néfazodone, verapamil, diltiazem
* Severe chronic liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The Primary efficacy measure is hospital mortality to day 28. | 28 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: LAURENT PAPAZIAN, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Papazian L, Roch A, Charles PE, Penot-Ragon C, Perrin G, Roulier P, Goutorbe P, Lefrant JY, Wiramus S, Jung B, Perbet S, Hernu R, Nau A, Baldesi O, Allardet-Servent J, Baumstarck K, Jouve E, Moussa M, Hraiech S, Guervilly C, Forel JM; STATIN-VAP Study Group. Effect of statin therapy on mortality in patients with ventilator-associated pneumonia: a randomized clinical trial. JAMA. 2013 Oct 23;310(16):1692-700. doi: 10.1001/jama.2013.280031. PMID 24108510